CLINICAL TRIAL: NCT03404713
Title: Evaluating the Feasibility of a Stepped-care Approach to Treating Adolescents With Binge and Loss of Control Eating
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant enrollment into stepped-care model was not feasible.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM20010755
Record Dates: First submitted 2018-01-03; First posted 2018-01-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity; Pediatric Obesity; Eating, Binge
Keywords: adolescence; adolescent; binge eating; loss-of-control eating; behavioral weight loss; weight management; acceptance commitment therapy; overweight; obesity
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity; Bulimia

STUDY DESIGN:
Intervention Model Description: Each eligible participant receives the same standard group treatment for the first four weeks. Early responders continue in that treatment for an additional 12 weeks. Early weak responders are assigned to a higher intensity individualized treatment for the next 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Behavioral Weight Loss (BWL) Treatment (Active Comparator): All participants will participate in 4 weeks of group based behavioral weight lost treatment in the intervention called Pathways to Health. Based on early treatment response (improvement in binge eating), participants will be assigned to either continue in this arm for the remaining 12 weeks of treatment (early strong responders) or be assigned to the 2nd arm of this study.
  Interventions: Behavioral: Pathways to Health
- Acceptance-Based Binge Eating Treatment (Experimental): After 4 weeks of standard BWL treatment, early weak responders will be assigned to individual acceptance-based treatment for the remaining 12 weeks of treatment.
  Interventions: Behavioral: Pathways to Health; Behavioral: Be4U

INTERVENTIONS:
Behavioral: Pathways to Health — Manualized sessions will follow an acceptance based behavioral weight loss treatment approach, including guided goal-setting and self-monitoring, identifying barriers and solutions, contingency management, stimulus control, dealing with setbacks and relapse prevention. Daily food and physical activity are logged and monitored. Parents learn strategies to support and facilitate their child's weight management via family-based change.
Behavioral: Be4U — This intervention is grounded in Cognitive Behavioral Therapy (CBT), Dialectical Behavioral Therapy (DBT), and Acceptance and Commitment Therapy (ACT). The core elements include regulating eating patterns, self-monitoring, developing openness to an acceptance perspective, fostering a willingness to accept distress, teaching defusion from distressing thoughts and feelings, practicing mindful awareness, fostering self-as-context, and directing patients towards clarifying and focusing on life values. Self-monitoring of eating behaviors and emotions are encouraged using a free app that facilitates electronic self-monitoring of eating patterns and symptoms. For participants who elect not to use this app, paper self-monitoring records are provided.
  Other Names: Acceptance-Based Binge Eating Intervention (ABBT)
  Arms: Acceptance-Based Binge Eating Treatment

SUMMARY:
There are limited evidence-based treatments for adolescents with binge eating and fewer specifically targeting adolescents with both binge eating and overweight/obesity. The existing research for adolescents with overweight/obesity and loss of control (LOC) eating supports a stepped-care model of treatment in which enhanced behavioral weight loss treatment is the first line of treatment followed by more intensive therapeutic treatment for individuals with remaining emotional eating difficulties. Thus, in this proposed study, the investigators will systematically develop a stepped-care protocol and manualized interventions for adolescents with LOC and binge eating behaviors. The investigators will then evaluate the feasibility and acceptability of the interventions in a pilot trial and gather preliminary outcome data to inform development of a subsequent randomized controlled trial.

DETAILED DESCRIPTION:
Binge eating affects a significant number of adolescents. Among adolescents seeking obesity treatment, rates of binge eating behavior range from 20-36%. Studies of non-treatment seeking adolescents have also identified high rates of binge eating, suggesting that this behavior is not exclusive to clinical samples. Moreover, as in adults, binge eating in youth is associated with numerous psychosocial problems, including depression, anxiety, low self-esteem, body dissatisfaction and weight concern.

Stepped-care models provide a lower intensity treatment and modify subsequent treatment intensity based on early treatment response. A stepped-care model would build upon the clinical treatment resources already established at the study site.

In this study, the investigators will conduct a small pilot of the stepped-care model. All participants will begin with the same initial treatment, an introductory behavioral weight loss group for parents and adolescents with abnormal weight gain and/or overweight/obesity. Early responders will continue in this treatment for an additional 12 weeks. Participants who show a weaker early response will be assigned to a higher intensity individualized treatment. All participants will receive 16 weeks of treatment.Assessments will occur at three time points: prior to intervention (baseline), mid-treatment (4 weeks), and end of treatment (16 weeks). The investigators will assess the feasibility, acceptability, and preliminary effectiveness of the stepped care approach. These data will inform the development of a subsequent RCT.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* Overweight (BMI ≥85% percentile for age and gender according to the CDC Growth Charts)
* Males and females ages 13 to 18 years
* Must endorse loss of control (LOC) eating
* Adolescent must reside with the primary participating caregiver who is also willing to participate in the study

Caregiver Inclusion Criteria:

* Participating caregiver must be at least 18 years of age
* Participating caregiver must reside with the adolescent
* Participating caregiver must be willing to participate in the standard intervention
* Participating caregiver may be another relative (i.e., grandparents) or legal guardian as long as he/she resides with the adolescent and has primary responsibility for the child.

Adolescent Exclusion Criteria:

* Non-English speaking
* Medical condition(s) that may be associated with unintentional weight change (e.g., hypothalamic injury, Prader Willi, or malignancy)
* Uncontrolled diabetes mellitus diagnosed by history or a fasting glucose ≥126 mg/dl (subjects with glucose intolerance or "prediabetes" will be eligible for study participation)
* Use of oral glucocorticoids, atypical antipsychotics, weight loss medications, diuretic medication or an investigational medication within 3 months of study participation
* Medical condition(s) that may be negatively impacted by exercise
* Psychiatric, cognitive, physical or developmental conditions that would impair the adolescent's ability to complete assessments, participate in a group, or conduct physical activity
* Reports of compensatory behaviors (i.e., vomiting, laxative, abuse, excessive exercise) in the past 3 months
* Current pregnancy or plan to become pregnant during study period
* Previous participation in Clinical Trials #(INSERT)
* Current participation in another weight loss program
* Personal history of weight loss surgery
* Weight in excess of 400 pounds
* Admission to a psychiatric hospital within the past year.

In addition, adolescents will be excluded from participation (and referred for further evaluation) based on the results of baseline psychological assessments under the following circumstances: 1) clinically significant depression, evidenced RCADS or or during screening / behavioral interview; 2) active suicidality as reported on surveys or during screening / behavioral interview; 3) clinically significant eating disorder based on assessments or during screening/behavioral interview.

Adolescents taking metformin, oral contraceptives, tricyclic antidepressants (TCAs), selective serotonin reuptake inhibitors (SSRIs), or stimulant medications may be eligible for participation; however, subjects must be on a stable dose of medication for at least 3 months prior to study participation.

Caregiver Exclusion Criteria:

* Non-English speaking
* Psychiatric, cognitive, physical or developmental conditions that would impair the parent's ability to respond to assessments or support adolescent's participation.

In the event that a participant is deemed eligible to participate based on initial criteria, but subsequently develops a condition listed for exclusion after participation in the study has begun, the investigative team will review the specific case to assess the impact of the newly discovered condition on the subject's ability to safely continue participation and the quality of the data that will be collected from the subject.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Change in objective and subjective binge and loss-of-control eating episodes as measured by the Eating Disorder Examination | Baseline, mid-treatment (4 weeks), and end of treatment (16 weeks)
  The overeating module of the Eating Disorder Examination (EDE) assesses frequency of adolescents' objective and subjective binge and loss-of-control eating episodes during the last 28 days. Change in frequency of these episodes from baseline will be assessed at 4 weeks and 16 weeks.

SECONDARY OUTCOMES:
Change in emotional eating as measured by the Emotional Eating Scale for Adolescents Questionnaire | Baseline, mid-treatment (4 weeks), and end of treatment (16 weeks)
  The Emotional Eating Scale for Adolescents Questionnaire (EES-C) measures an adolescent's desire to eat as a means of coping with emotions. Change in emotional eating from baseline will be assessed at 4 weeks and 16 weeks.
Change in anxiety and depressive symptoms as measured by the Revised Child Anxiety and Depression scales | Baseline, mid-treatment (4 weeks), and end of treatment (16 weeks)
  The Revised Child Anxiety and Depression scales assess adolescent mood, specifically anxiety and depressive symptoms; both adolescent self-report and caregiver report will be collected. Change in these measures from baseline will be assessed at 4 weeks and 16 weeks.
Change in self-esteem as measured by the Rosenberg Self-Esteem Scale | Baseline, mid-treatment (4 weeks), and end of treatment (16 weeks)
  The Rosenberg Self-Esteem Scale (RSES) measures an adolescent's global self-reported self-worth. Change in self-esteem from baseline will be assessed at 4 weeks and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel W Gow, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States